CLINICAL TRIAL: NCT04111991
Title: Effectiveness of a Psychological Intervention for Children With Post-concussion Syndrome
Brief Title: Concussion Symptom Treatment and Education Program (C-STEP) in Post-Concussion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sean Rose (Other)
Collaborators: Nationwide Children's Hospital (Other); Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Sean Rose, Assistant Professor of Pediatrics, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000529
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-03

CONDITIONS: Post-Concussion Syndrome
Keywords: Behavior Therapy, Cognitive; Post-Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Usual care in the NCH Complex Concussion Clinic
  Interventions: Behavioral: Usual Care
- Usual Care + C-STEP (Experimental): Usual care in the NCH Complex Concussion Clinic, plus 4 weekly sessions of C-STEP
  Interventions: Behavioral: Usual Care; Behavioral: C-STEP (Cognitive Behavioral Therapy)

INTERVENTIONS:
Behavioral: Usual Care — Usual care in the NCH in the Complex Concussion Clinic involves assessment and treatment with a neurologist for medical management of concussion, weekly sessions with an athletic trainer for exercise therapy, and physical therapy sessions depending on need
Behavioral: C-STEP (Cognitive Behavioral Therapy) — The C-STEP intervention involves 4 primary components: psychoeducation, activity management, sleep hygiene, and relaxation training
  Arms: Usual Care + C-STEP

SUMMARY:
This prospective randomized intervention study aims to determine if the Concussion Symptom Treatment Program (C-STEP), a cognitive behavioral therapy, improves outcomes for children with post-concussion syndrome.

DETAILED DESCRIPTION:
This prospective randomized intervention study aims to determine if C-STEP improves outcomes for children with post-concussion syndrome. Forty children with post-concussion syndrome referred to the Nationwide Children's Hospital (NCH) Complex Concussion Clinic will be randomized to receive either usual care in the NCH Complex Concussion Clinic (comparison) or usual care in the NCH Complex Concussion Clinic plus four weekly sessions of C-STEP (treatment).

C-STEP has been developed for patients with post-concussion syndrome. The CBT intervention involves 4 primary components: psychoeducation, activity management, sleep hygiene, and relaxation training (adapted from McNally et al., 2018). Psychoeducation involves providing patients and families with information about typical concussion symptoms and recovery, the role of non-injury/psychological factors in post-concussion syndrome, and information about the mind-body connection. Activity management involves setting specific goals to achieve a return to normal daily activities such as school attendance, schoolwork completion, household activities, and participating in social/leisure activities. The sleep hygiene component involves providing individualized recommendations to promote healthy sleep habits such as eliminating naps, keeping a consistent sleep schedule, turning off electronics at bedtime, or other needed modifications. Finally, relaxation training involves teaching specific evidence-based strategies for relaxation and coping with stress such as diaphragmatic breathing and progressive muscle relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Children age 10-17 years or adults age 18 years (total age range 10-18) at the time of the enrollment visit
* Diagnosed concussion occurring between 1 month and 12 months prior to the enrollment visit
* Endorsing at least 2 symptoms on the SCAT-5 symptom checklist
* Intent to participate in the full CCC treatment program (including exercise visits once per week)

Exclusion Criteria:

* Adults unable to consent, Prisoners, Females currently known to be pregnant, Non-English speaking patient
* Anticipated inability to complete surveys or other study procedures (due to cognitive or other disability)
* Anticipated inability to complete a brain MRI (due to claustrophobia, implanted hardware or other contraindications)
* Pre-injury severe mental illness (defined as inpatient psychiatric hospitalization, suicide attempt, history of psychotic symptoms, or bipolar disorder)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Sport Concussion Assessment Tool- Fifth Edition (SCAT-5) Concussion Symptoms | Day 0 to Day 35
  This is a 22-item self and parent-reported list of common concussion symptoms filled out on a 0-6 Likert scale. Scores range from 0 to 122. Higher scores are indicative of worse concussion symptoms.
Change Pediatric Quality of Life Inventory, Version 4.0 (PedsQL) | Day 0 to Day 35
  This is a 23-item self and parent-reported quality of life metric. Each item is rated on a scale of 0-4. Scores range from 0-100 for each subscale (Physical Functioning; Emotional Functioning; Social Functioning; School Functioning) and for the total score. Higher scores are indicative of better quality of life.

SECONDARY OUTCOMES:
Change in Brain Connectivity | Day 0 to Day 35
  An advanced neuroimaging protocol will measure brain tissue volume, microstructure, and function.
Change in Auditory Attention and Working Memory | Day 0 to Day 35
  The digit span forwards and backwards subtest from Wechsler Individual Scales of Intelligence, fifth edition (WISC-V) (age 12-16) or Wechsler Adult Intelligence Scales, fourth edition (WAIS-IV) (age 17-18) will test auditory attention and working memory. Age-normed scaled scores (range 1-19, higher is better performance) will be calculated for process scores of Digits Forward and Digits backward.
Change in Processing Speed | Day 0 to Day 35
  The processing speed index, which consists of the Coding and Symbol Search subtests from the from WISC-V (age 12-16) or WAIS-IV (age 17-18) will test processing speed. Age-normed scaled scores (range 1-19, higher is better performance) will be calculated for Coding and Symbol Search subtests. Scaled scores for these will be summed and used to calculate the Processing Speed Index standard score (range 45-155, higher is better performance).
Change in Phonemic Verbal Fluency | Day 0 to Day 35
  The Phonemic Verbal Fluency (letter fluency) subtest from the Delis Kaplan Executive Function Scales (DKEFS) will test executive functioning and phonemic verbal fluency. Age-normed scaled scores (range 1-19, higher is better performance) will be calculated for the phonemic fluency subtest.
Change in Cognitive Flexibility | Day 0 to Day 35
  The Letter Number Sequencing subtest from from DKEFS will test cognitive flexiblity. Age-normed scaled scores (range 1-19, higher is better performance) will be calculated for the number sequencing and letter-number sequencing trials.
Change in Verbal Memory | Day 0 to Day 35
  The Lists (immediate, delayed, and recognition) subtest from the Child and Adolescent Memory Profile (ChAMP) tests verbal memory. Age-normed scaled scores (range 1-19, higher is better performance) will be calculated for Lists, Lists Delayed, and Lists recognition subtests.
Change in Performance Validity | Day 0 to Day 35
  The Medical Symptom Validity Test- (MSVT) will test effort/performance validity. Percentage scores for immediate recognition, delayed recognition, consistency, paired associates, and free recalls will be calculated. Performance will be classified as Pass vs. Fail.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Rose, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No